CLINICAL TRIAL: NCT01300949
Title: Validation and Reproducibility of Spaeth/Richman Contrast Sensitivity Test
Brief Title: Spaeth/Richman Contrast Sensitivity Test
Acronym: SPARCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, George L. Spaeth MD, Principal Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-998
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Results first posted 2018-11-08 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Glaucoma
Keywords: Contrast Sensitivity; Pelli-Robson Test
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Contrast sensitivity, another means of testing vision, will be measured two ways for each participant. One method uses the Pelli-Robson Contrast Sensitivity Chart which is mounted on the wall, the other method uses a new computerized program called Spaeth/Richman Contrast Sensitivity Test also known as SPARCS.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glaucoma (Active Comparator): 154 glaucoma, ocular hypertension and glaucoma suspect patients will have contrast sensitivity measured by Spaeth/Richman Contrast Sensitivity Test (SPARCS) and Pelli-Robson Contrast Sensitivity Chart.
  Interventions: Diagnostic Test: Spaeth/Richman Contrast Sensitivity Test; Diagnostic Test: Pelli-Robson Contrast Sensitivity Chart
- Controls (Active Comparator): 125 patients with no eye diseases will have contrast sensitivity measured by Spaeth/Richman Contrast Sensitivity Test (SPARCS) and Pelli-Robson Contrast Sensitivity Chart. This included patients with refractive errors (needing glasses) and nuclear sclerosis (cataract).
  Interventions: Diagnostic Test: Spaeth/Richman Contrast Sensitivity Test; Diagnostic Test: Pelli-Robson Contrast Sensitivity Chart
- Age-Related Macular Degeneration (ARMD) (Active Comparator): 35 retina patients with age-related macular degeneration (ARMD) will have contrast sensitivity measured by Spaeth/Richman Contrast Sensitivity Test (SPARCS) and Pelli-Robson Contrast Sensitivity Chart.
  Interventions: Diagnostic Test: Spaeth/Richman Contrast Sensitivity Test; Diagnostic Test: Pelli-Robson Contrast Sensitivity Chart

INTERVENTIONS:
Diagnostic Test: Spaeth/Richman Contrast Sensitivity Test — internet based computerized contrast sensitivity test measuring central and peripheral vision using black and white stripes that decrease in contrast by fading to a white background.
  Other Names: SPARCS
Diagnostic Test: Pelli-Robson Contrast Sensitivity Chart — wall chart contrast sensitivity test measuring central vision using black letters that decrease in contrast by fading to a white background.

SUMMARY:
The Spaeth-Richman Contrast Sensitivity (SPARCS) test is a new method of assessing contrast sensitivity. The test, another way to measure vision, is performed on any standard computer with internet access. Patients will be tested with SPARCS and with the standard Pelli-Robson contrast test.

DETAILED DESCRIPTION:
Contrast Sensitivity is another way to test vision. It uses black on a white background and minimally decreases the black (grey) until it blends with the white. The least amount of contrast (faint grey) seen translates into amount of vision. This new method of determining contrast sensitivity uses black and white vertical bars and does not require recognizing letters in the alphabet. It tests various areas of the visual field and central vision. The test takes approximately 3 minutes per eye.

Pelli-Robson is a commonly used contrast sensitivity test that uses black letters on a white background. The letter size stays the same, only the amount of black changes, becoming greyer, making letters hard to see. The test takes approximately 1 minute per eye.

Hypothesis: A method of determining contrast sensitivity that does not require letter recognition (as does the Pelli-Robson test) eliminates the barriers of literacy and pattern recognition, to permit a more valid determination of contrast sensitivity.

Patients will perform SPARCS and Pelli-Robson twice; once each with two separate observers for reproducibility and intra-observer reliability. The order of testing will be randomized to SPARCS, Pelli, Pelli, SPARCS or Pelli, SPARCS, SPARCS, Pelli.

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs of age and older
* able to provide fully informed consent

  70 controls (patients with no ocular disease affecting visual acuity or visual function), 10 from each decade of life: 20-30, 30-40, 40-50, 50-60, 60-70, 70-80, 80+.

  105 patients with ocular hypertension or any type of glaucoma (15 subjects per age decade). Glaucoma patients will not have macular degeneration or visual acuity affected by any function other than glaucoma.

  40 patients with macular degeneration: 10 with visual acuity 20/40 or better, 10 with visual acuity between 20/40 and 20/60, 10between 20/100 and 20/400, and 10 with 20/400 or worse.

  40 patients with cataracts: 10 with lens opacity 1+nuclear sclerosis, 10 with 2 + nuclear sclerosis, 10 with 3 + nuclear sclerosis, 10 with 4 + nuclear sclerosis.

  60 patients with refractive error: 10 with myopia -5 diopters or greater, 10 with myopia between -5 and -2.5, 10 with myopia between -2.5 and -0.5, 10 with myopia between -0.5 and 0.5, 10 with myopia between 0.5 and 2.5, and 10 with myopia > 2.5.

Exclusion Criteria:

* any other diseases affecting visual acuity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George L Spaeth, MD, Principal Investigator — Glaucoma Service, Wills Eye Institute
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Multiple manuscripts have been published.

REFERENCES:
- [Result] Richman J, Zangalli C, Lu L, Wizov SS, Spaeth E, Spaeth GL. The Spaeth/Richman contrast sensitivity test (SPARCS): design, reproducibility and ability to identify patients with glaucoma. Br J Ophthalmol. 2015 Jan;99(1):16-20. doi: 10.1136/bjophthalmol-2014-305223. Epub 2014 Jul 22. PMID 25053760
- [Result] Faria BM, Duman F, Zheng CX, Waisbourd M, Gupta L, Ali M, Zangalli C, Lu L, Wizov SS, Spaeth E, Richman J, Spaeth GL. EVALUATING CONTRAST SENSITIVITY IN AGE-RELATED MACULAR DEGENERATION USING A NOVEL COMPUTER-BASED TEST, THE SPAETH/RICHMAN CONTRAST SENSITIVITY TEST. Retina. 2015 Jul;35(7):1465-73. doi: 10.1097/IAE.0000000000000474. PMID 25658175
- [Result] Sun Y, Erdem E, Lyu A, Zangalli C, Wizov SS, Lo D, Spaeth EE, Richman J, Spaeth GL. The SPARCS: a novel assessment of contrast sensitivity and its reliability in patients with corrected refractive error. Br J Ophthalmol. 2016 Oct;100(10):1421-6. doi: 10.1136/bjophthalmol-2015-307378. Epub 2016 Jan 12. PMID 26758536
- [Result] Gupta L, Cvintal V, Delvadia R, Sun Y, Erdem E, Zangalli C, Lu L, Wizov SS, Richman J, Spaeth E, Spaeth GL. SPARCS and Pelli-Robson contrast sensitivity testing in normal controls and patients with cataract. Eye (Lond). 2017 May;31(5):753-761. doi: 10.1038/eye.2016.319. Epub 2017 Jan 20. PMID 28106888

RESULTS

PARTICIPANT FLOW:
Groups:
- Glaucoma: 154 glaucoma, ocular hypertension and glaucoma suspect patients
- Controls: 125 patients with no eye diseases. This included patients with refractive errors (needing glasses) and nuclear sclerosis (cataract).
- Age-Related Macular Degeneration (ARMD): 35 retina patients with age-related macular degeneration (ARMD)
Period: Overall Study
Arm/Group | Glaucoma | Controls | Age-Related Macular Degeneration (ARMD)
Started | 154 | 125 | 35
Completed | 154 | 125 | 35
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glaucoma | Controls | Age-Related Macular Degeneration (ARMD) | Total
Number analyzed (Participants) | 154 | 125 | 35 | 314
Age, Continuous [Mean (Full Range); unit: years] | 68 [19 to 98] | 49 [20 to 83] | 81 [74 to 88] | 62 [19 to 98]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 65 | 17 | 162
  Male | 74 | 60 | 18 | 152
Region of Enrollment [Number; unit: participants]
  United States | 154 | 125 | 35 | 314

OUTCOME MEASURES:

1. Primary Outcome: Contrast Sensitivity, Another Means of Testing Vision
Description: Contrast Sensitivity, a vision measurement, is performed with the Spaeth Richmond Contrast Sensitivity (SPARCS) test. This is a computerized measurement of vision in the central and peripheral fields using black and white stripes. Black stripes decrease in contrast becoming fainter and harder to see until they blend with the white background. Measurements are assessed in five areas of the visual field . Test results are reported for each area ranging from 0 to 20 (0 means can't see stripes; 20 means sees all stripes). Results from all 5 areas are added making the total SPARCS score range 0 - 100 where 0 means poor vision and 100 means best vision. The test takes an average of 3 minutes per eye. The eye not being tested is covered with a patch.
Time Frame: duration of 1 eye exam, approximately 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Glaucoma: 154 glaucoma, ocular hypertension and glaucoma suspect patients
  Spaeth/Richman Contrast Sensitivity Test: internet based computerized contrast sensitivity test measuring central and peripheral vision using black and white stripes
  Pelli-Robson Contrast Sensitivity Chart: chart measuring central vision with black letters fading to white on a white background
- Controls: 125 patients with no eye diseases. This included patients with refractive errors (needing glasses) and nuclear sclerosis (cataract).
  Spaeth/Richman Contrast Sensitivity Test: internet based computerized contrast sensitivity test measuring central and peripheral vision using black and white stripes
  Pelli-Robson Contrast Sensitivity Chart: chart measuring central vision with black letters fading to white on a white background
- Age-Related Macular Degeneration (ARMD): 35 retina patients with age-related macular degeneration (ARMD)
  Spaeth/Richman Contrast Sensitivity Test: internet based computerized contrast sensitivity test measuring central and peripheral vision using black and white stripes
  Pelli-Robson Contrast Sensitivity Chart: chart measuring central vision with black letters fading to white on a white background
Arm/Group | Glaucoma | Controls | Age-Related Macular Degeneration (ARMD)
Number analyzed (Participants) | 154 | 125 | 35
units on a scale | 59.4 (15.3) | 74.4 (5.0) | 53.9 (19)

ADVERSE EVENTS:
Time Frame: duration of 1 eye exam, approximately 1 hour
Arm/Group | Glaucoma | Controls | Age-Related Macular Degeneration (ARMD)
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/125 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/125 | 0/35
Other Adverse Events (participants affected / at risk) | 0/154 | 0/125 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No